CLINICAL TRIAL: NCT02762201
Title: Clinical Evaluation of Therapeutic Efficiency of Implant-secured Removable Partial Denture: A Randomized, Controlled, Prospective Multicentric Study.
Brief Title: Clinical Evaluation of Implant-secured Removable Partial Denture
Acronym: PASI-PAC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor and principal investigator decision
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-726
Record Dates: First submitted 2016-05-03; First posted 2016-05-04 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Tooth Loss
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PASI (Experimental): PASI dental prosthesis delivery
  Interventions: Procedure: PASI
- PAC (Active Comparator): PAC dental prosthesis delivery
  Interventions: Procedure: PAC

INTERVENTIONS:
Procedure: PASI — Implant-secured removable partial denture will be delivered in 2 large steps: implant delivery followed by denture delivery.
  * Implant delivery will take 4 dental consultations : a pre-implant study at Day14 after inclusion, the surgical implant insertion at D28 after inclusion, stitches removal at D35 after inclusion, and finally functional implant delivery between 3 or 6 month after surgery (to allow implant osteointegration).
  * Denture delivery will take 6 weekly dental consultations between Week 3 and Week 8 after the functional implant delivery.
  Arms: PASI
Procedure: PAC — Metalic standard removable partial denture, the standard treatment, will be delivered in 4 steps at Day 7, D14, D21, D28 after inclusion, as classically.
  Arms: PAC

SUMMARY:
This study aims to compare the therapeutic efficiency of implant-secured removable partial denture (PASI) with the therapeutic efficiency of the metalic standard removable partial denture (PAC) in the treatment of intermediate extended-gap (4 adjacent teeth). The therapeutic efficiency will be assessed by the 5 years-prosthetic success rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least a 4 to 6 adjacent teeth intermediate extended-gap (excluding wisdom teeth) in the upper or lower jaw.
* Patients with at least 4 conservable teeth by dental arch, without major occlusal trouble.
* Patients with healthy periodontium, allowing metalic standard removable partial denture delivery : bleeding on periodontal probing for a duration less than 30 seconds, Osteolysis of the alveolar ridge less or equal to 50%, attachment loss less or equal to 5mm
* Patients with a sufficient bone volume for implant placement, without prior bone supply.

Exclusion Criteria:

* Patients with general counter-indications for implant placement.
* Patients suffering from a titanium allergy.
* Patients with an insufficient oral and dental hygiene - Patients smoking ten or more cigarettes per day.
* Patients with teeth extended-gap, which could be corrected by a fixed tooth-supported denture.
* Patient with an insufficient available bite level to deliver an attachment system (< 7mm).
* Patients with a severe generalized chronic periodontitis , an aggressive periodontitis or a periodontitis unresponsive to treatment.
* Women who have reported to be pregnant.
* Patients deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-05-16 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2019-06-06 (Actual)

PRIMARY OUTCOMES:
prosthetic success rate | 5 years after prosthesis delivery

SECONDARY OUTCOMES:
prosthetic success rate | 6 months, 1 year, 2 years, 3 years and 4 years after prosthesis delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No